CLINICAL TRIAL: NCT06070350
Title: Massive Transfusion in Children: a Platform RCT of Whole Blood Compared to Component Therapy and Tranexamic Acid to Placebo in Life-threatening Traumatic Bleeding
Brief Title: Massive Transfusion in Children-2: A Trial Examining Life Threatening Hemorrhage in Children
Acronym: MATIC-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Philip Spinella (Other)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Philip Spinella, Professor of Surgery and Critical Care Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MATIC-002
Record Dates: First submitted 2023-09-27; First posted 2023-10-06 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Hemorrhagic Shock; Trauma Injury
Keywords: Children; Pediatrics; Transfusion
MeSH Terms: conditions — Shock, Hemorrhagic; Accidental Injuries | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: MATIC-2 is a Bayesian, randomized, multicenter, adaptive platform phase III trial to examine the effectiveness and safety of LTOWB versus CT and TXA vs placebo in 1000 children at minimum 20 US high volume academic pediatric trauma centers. Mechanisms of Trauma induced Coagulopathy (TIC) and resuscitation effects will also be investigated. The trial will stratify pediatric trauma centers based on their reported Massive Transfusion Protocol (MTP) volume and then randomize them into four treatment combinations. After an initial enrollment phase, treatment sites will cross over to ensure that all treatments are tested across every site, eliminating biases by the time of the first interim analysis.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The University of Pittsburgh Medical Center Investigational Research Pharmacy will provide each site the placebo and TXA. The research pharmacy at each site will draw the dose syringes. They will be blinded with a label indicating either drug A or B, and the pharmacy will log which patients received TXA or placebo, with all drugs labeled as investigational products.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (LTOWB+TXA) (Other): Concurrent administration of LTOWB and TXA
  Interventions: Biological: Low Titer Group O Whole Blood (LTOWB); Drug: Tranexamic Acid (TXA)
- Group 2 (LTOWB+Placebo) (Other): Concurrent administration of LTOWB and Placebo
  Interventions: Biological: Low Titer Group O Whole Blood (LTOWB); Drug: Placebo
- Group 3 (CT+TXA) (Other): Concurrent administration of CT and TXA
  Interventions: Drug: Tranexamic Acid (TXA); Biological: Component Therapy (CT)
- Group 4 (CT+Placebo) (Other): Concurrent administration of CT and Placebo
  Interventions: Drug: Placebo; Biological: Component Therapy (CT)

INTERVENTIONS:
Biological: Low Titer Group O Whole Blood (LTOWB) — LTOWB is whole blood from group O donors with low titer (<200) anti-A and anti-B antibodies. Up to 8 units of LTOWB will be allowed unless local clinical practice allows for a higher maximum dose.
  Arms: Group 1 (LTOWB+TXA); Group 2 (LTOWB+Placebo)
Drug: Placebo — Placebo will be provided to the research pharmacy at each of the clinical sites
  Arms: Group 2 (LTOWB+Placebo); Group 4 (CT+Placebo)
Drug: Tranexamic Acid (TXA) — TXA is a synthetic lysine analog that competitively inhibit activation of plasminogen, thereby decreasing the conversion of plasminogen to plasmin, preventing degradation of fibrin's matrix structure. Dose is 25mg/kg IV or IO (maximum 2 grams).
  Arms: Group 1 (LTOWB+TXA); Group 3 (CT+TXA)
Biological: Component Therapy (CT) — Component Therapy (CT) will be RBCs, plasma and platelet units in a 1:1:1 unit ratio. This will be given with Placebo
  Arms: Group 3 (CT+TXA); Group 4 (CT+Placebo)

SUMMARY:
The MATIC-2 is a multicenter clinical trial enrolling children who are less than 18 years of age with hemorrhagic shock potentially needing significant blood transfusion.

The primary objective of the clinical trial is to determine the effectiveness of Low Titer Group O Whole Blood (LTOWB) compared to component therapy (CT), and Tranexamic Acid (TXA) compared to placebo in decreasing 24-hour all-cause mortality in children with traumatic life threatening hemorrhage.

DETAILED DESCRIPTION:
The MATIC-2 trial is a Bayesian, randomized, multicenter, adaptive platform phase III trial. The trial will include injured children with hemorrhagic shock anticipated to require massive blood transfusion, who will be randomized to receive either LTOWB or CT and Tranexamic Acid or placebo.

The study investigators hypothesize that the use of LTOWB is non-inferior and/or superior for 24-hour mortality and that LTOWB does not increase the risk of adverse events or outcomes, such as thrombotic events, compared to CT.

The investigators also hypothesize that the use of TXA is superior for 24-hour mortality and does not increase the risk of adverse events or outcomes, such as thrombotic events, compared to placebo.

Objectives:

The primary objectives are to:

1. Determine the effectiveness of LTOWB to reduce all-cause 24-hour mortality compared to CT in children with traumatic life-threatening hemorrhage.
2. Determine the effectiveness of TXA to reduce all-cause 24-hour mortality compared to placebo in children with traumatic life-threatening hemorrhage.

Secondary objectives are to determine the effectiveness and safety of LTOWB and TXA to improve secondary and exploratory outcomes (or endpoints) in children with traumatic life-threatening hemorrhage.

Safety objectives are to determine the effect of LTOWB and TXA on safety related outcomes/endpoints. The safety outcomes include:

1. Acute kidney injury
2. Acute respiratory distress syndrome
3. Arrhythmia
4. Abdominal compartment syndrome
5. Bleeding after hemostasis requiring intervention
6. Myocardial infarction
7. Pneumonia
8. Sepsis
9. Stroke
10. Seizure
11. Thrombotic events (arterial or venous)
12. Urinary Tract Infection
13. Alloimmunization in Rh negative female recipients of Rh+ LTOWB or RBC's
14. Organ failure (as determined by PELOD-2 score)

Mechanistic Objectives are to:

1. Define trauma induced coagulopathy (TIC) according to measures of shock, hemostasis, and endothelial and immune function.
2. To determine if measures of shock, endothelial, immune, and hemostasis function upon admission (TIC endotype) predicts which hemostatic resuscitation therapies or combinations of therapies (LTOWB, CT, LTOWB + TXA, CT+TXA) for each study group improves outcomes without increasing the risk of adverse events.
3. To determine the mechanisms of how hemostatic resuscitation therapies or combinations of therapies (LTOWB, CT, LTOWB + TXA, CT+TXA) improve TIC endotypes and outcomes.

Pharmacokinetic objectives are to evaluate the PK and PD properties of TXA in a population of children with life-threatening traumatic bleeding.

ELIGIBILITY:
General Inclusion Criteria:

1. Children, defined as less than estimated18 years of age with traumatic injury
2. MTP activation for confirmed or suspected active life-threatening traumatic bleeding

AND

Confirmed or suspected active life-threatening traumatic bleeding with at least 2 of 3 of the following criteria:

1. Hypotension for age (< 5% tile)
2. Tachycardia for age (>95th % tile)
3. Traumatic injury with exam findings consistent with severe bleeding (e.g., penetrating injury, hemothorax, distended abdomen with bruising, amputation of limb).

General Exclusion Criteria:

1. Patient with devastating traumatic brain injury not expected to survive due to magnitude of injury (example: Transhemispheric gunshot wound with signs of herniation, GCS score of 3 with fixed and dilated pupils)
2. MTP activated but no blood products given
3. Patients who required an ED thoracotomy or received more than 5 consecutive minutes of cardiopulmonary resuscitation (prior to receiving randomized blood products)
4. Patients who are known or suspected to be pregnant on clinical examination
5. Known prisoners as defined in protocol
6. Known ward of the state
7. Isolated hanging, drowning or burns
8. Previous enrollment in MATIC-2
9. Prior study opt-out with bracelet

Exclusion Criteria for the TXA/Placebo Domain

1. Prehospital or pre-enrollment use of TXA
2. Greater than 3 hours since time of injury
3. History of seizure after the injury event
4. Known allergy or hypersensitivity reaction to TXA

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
24 hours all cause mortality | 24 hours

SECONDARY OUTCOMES:
6-hour, 72-hour and 28-day survival | 6, 72 hours and 28 days
  Cumulative survival over time through 28 days post-enrollment: includes 6-hour, 72-hour and 28-day survival.
24 hours total blood product transfusion volumes | 24 hours
  Total blood product transfusion in 24 hours after enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Philip C Spinella, MD, Principal Investigator — Univesrity of Pittsburgh
Locations (23):
- United States (23):
  - University of Arizona, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of California Davis, Sacramento, California
  - Children's National Hospital, Washington D.C., District of Columbia
  - Emory University-Arthur M. Blank Hospital, Atlanta, Georgia
  - Emory University-Scottish Rite Hospital, Atlanta, Georgia
  - Tulane School of Medicine, New Orleans, Louisiana
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University of St. Louis, St Louis, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - Wake Forest University Health Sciences, Wake Forest, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - LeBonheur Children's Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Children's Memorial Hermann Hospital, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Washington Harborview, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared 5 years after the trial has been published. The trial database will be shared to those who request the data and agree to collaborate with the principal investigators for the additional analyses.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Petersen EM, Fisher AD, April MD, Yazer MH, Braverman MA, Borgman MA, Schauer SG. The effect of the proportion of low-titer O whole blood for resuscitation in pediatric trauma patients on 6-, 12- and 24-hour survival. J Trauma Acute Care Surg. 2025 Apr 1;98(4):587-592. doi: 10.1097/TA.0000000000004564. Epub 2025 Feb 3. PMID 39898869